CLINICAL TRIAL: NCT05211700
Title: Socio-Clinical Factors Associated With Self-Management and Patient Activation in Parkinson's Disease
Brief Title: Socio-Clinical Factors Associated With Self-Management in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: University of Haifa (Other)
Collaborators: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Galit Yogev-Seligmann, Prinicipal Investigator, University of Haifa
Other Study IDs: 0067-19-RMB
Record Dates: First submitted 2021-12-30; First posted 2022-01-27 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is an observational study, there is no intervention in this study. — There is no intervention in this study

SUMMARY:
Self-management focuses on the behaviors that people with chronic disease use in order to maintain and improve their health and well-being and includes aspects such as medical and lifestyle management. Parkinson's disease (PD) is a chronic, progressive, incurable neurodegenerative disorder that affects motor and non-motor function. Engagement in self-management behaviors and high activation may be effective tools in fighting the long-lasting burden of the disease. The goal of the current study was to explore socio-clinical factors that associate with specific self-management behaviors and patient activation among patients with Parkinson's disease. PwP were recruited from the Movement Disorders Institute, Department of Neurology, Rambam Health Care Campus. Eligible patients were assessed for cognitive status and filled questionnaires regarding socio-clinical factors included age, gender, severity of motor and non -motor symptoms, family and social support. Data about the comorbidities were retrieved from electronic medical records

DETAILED DESCRIPTION:
n Parkinson's disease (PD), implementation of self-management strategies together with high patient activation may be an effective tool in fighting the long-lasting burden of the disease, but little is known about its determinant.

The aims of this study, conducted among patients with PD are to (1) test the association between socio-clinical factors that includes age, gender, cognitive status, comorbidities, disease severity (motor and non-motor symptoms) and social support and SMBs including utilization of rehabilitative treatments (an aspect of medical management), physical activity (an aspects of lifestyle management), and patient activation, and (2) to develop predictive model for each of these three aspects of SMB, based on socio-clinical factors that includes age, gender, cognitive status, comorbidities, disease severity (motor and non-motor symptoms) and social support.

A cross-sectional study of 100 patients that attend a Movement Disorder Clinic with PD will be conducted. Participation will include one evaluation session of approximately 90 minutes. Information about socio-clinical characteristics and self-management behaviors will be collected using demographic questionnaires, standard questionnaires and from electronic medical records. Regression model will test the association between sociodemographic characteristics and self-management behaviors and patient activation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD
* Age > 18

Exclusion Criteria:

• Mini Mental State Exam<20

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PD who are treated in the Movement Disorders Institute, Department of Neurology, Rambam Health Care Campus.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Patient's Activation Measure (PAM-13®️, Insignia Health) | through study completion, an average of 1 year
  Patient Activation Measure (PAM) score. Patient activation' describes the skills, confidence and knowledge a person has in managing her/his own health and health care.
  It consists of 13 statements rated on a four-point Likert scale of level of agreement. The PAM-13 score is transformed into a 0-100 continuous scale according to a licensed conversion table (Insignia Health)
International Physical Activity Questionnaire- IPAQ-SHORT | through study completion, an average of 1 year
  This questionnaire asks individuals to assess the number of days and amount of time they spent in the last 7 days in four categories: 1) vigorous activity (heavy lifting, aerobics, fast bicycling), 2) moderate activity (light lifting, moderate bicycling), 3) walking (at least 10 minutes), 4) sitting (watching TV, reading). Total physical activity is calculated as the sum of Walking + Moderate + Vigorous metabolic equivalent (MET) minutes/week scores.
Utilization of rehabilitative treatments | Through study completion, an average of 1 year
  Participants reported about whether and how frequently they utilize physical therapy, occupational therapy, and speech and language pathology treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Galit Yogev-Seligmann, Haifa, Please Select..., Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Duvdevani M, Yogev-Seligmann G, Schlesinger I, Nassar M, Erich I, Hadad R, Kafri M. Association of health behaviors with function and health-related quality of life among patients with Parkinson's disease. Isr J Health Policy Res. 2024 Jan 3;13(1):2. doi: 10.1186/s13584-023-00588-3. PMID 38173041